CLINICAL TRIAL: NCT00487799
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study of Ularitide in the Treatment of Subjects With Acute Decompensated Heart Failure
Brief Title: A Study of Ularitide in the Treatment of Subjects With Acute Decompensated Heart Failure
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Facet no longer has ownership of ularitide.
Sponsor: Facet Biotech (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ularitide-1503
Record Dates: First submitted 2007-06-15; First posted 2007-06-19 (Estimated); Last update posted 2009-07-20 (Estimated); Status verified 2009-07

CONDITIONS: Heart Failure, Congestive
Keywords: Acute Decompensated Heart Failure; ADHF; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Ularitide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Ularitide

SUMMARY:
To determine the maximum tolerated dose (MTD) of ularitide in the treatment of subjects hospitalized with symptomatic acute decompensated heart failure (ADHF).

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for inclusion, subjects must meet all of the following criteria:

* Males and females who are 18 years or older.
* Unplanned hospitalization for ADHF.
* Randomization should occur as soon as possible from presentation to emergency department or hospital for ADHF up to 24 hours from admission.
* Dyspnea at rest as assessed by the subject not more than 1 hour prior to randomization. Subjects must have the ability to interpret and report self-assessed dyspnea.
* At least 1 of the following 2 criteria:

  1. Prior medical history of CHF (eg, prior hospitalization for CHF or left ventricular ejection fraction <40%, as determined by transthoracic echocardiography at the time of screening or previously determined and documented in the patient's chart as follows):

     * Within the previous 6 months in subjects with unstable symptoms, or
     * Within the previous 12 months in subjects with stable symptoms.
  2. Clinical evidence (at screening) of heart failure, including abnormal jugular venous pressure (JVP) (eg, >8 cm above the clavicle, assessed at 45°angle), rales or crackles more than a third above bases, or 2+ lower extremity edema.
* On optimal background therapy for ADHF (as determined by the investigator); subjects are required to have received, at a minimum, at least 1 hour of oxygen supplementation and at least one dose of IV furosemide at a minimum dose of 40 mg with the last bolus being delivered >2 hours before study drug administration is initiated (or another diuretic at a comparable dose; eg, 2 mg bumetanide or 20 mg torsemide, with the last bolus being delivered >4 hours before study drug administration is initiated.
* If subject received IV opiate, the last dose must have been >3 hours before administration of study drug.
* Women of childbearing potential must have a negative pregnancy test prior to being randomized in the study. Women and men of reproductive potential will agree to utilize effective contraception during the entire treatment period and for 1 month after receiving the last dose of ularitide or placebo.
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations).

Exclusion Criteria:

Any subject will be ineligible for this study if any one of the following criteria is met:

* Breathing rate <18 breaths per minute (measured during 60 seconds).
* A systolic blood pressure (SBP) <110 mmHg or >180 mmHg within an hour before randomization, or SBP <120 mmHg for subjects receiving IV inotropics or vasodilators. A SBP <90 mmHg in two successive measurements within 30 minutes before randomization. (Subjects on baseline IV inotropes or vasodilators must be on a stable dose for ³3 hours prior to randomization.)
* BNP <400 pg/mL or NT?pro-BNP <1200 pg/mL anytime from initial presentation to hospital to time of randomization.
* Use of IV contrast material within 48 hours before infusion of study drug.
* History of central or peripheral neurological ischemic disorder (stroke, etc.).
* Active myocarditis, obstructive hypertrophic cardiomyopathy, congenital heart disease, restrictive cardiomyopathy, constrictive pericarditis, severe aortic stenosis, uncorrected primary valvular disease, or significant obstructive valve disease.
* Acute decompensated heart failure associated with endocrine (eg, thyroid storm), metabolic, or drug-related toxicity.
* Elevation of serum creatinine?kinase myocardial band (CK?MB) or cardiac troponin (Troponin I) >2 times the upper limit of normal within 6 hours prior to randomization.
* Active, ongoing myocardial ischemia, hospitalization for acute myocardial infarction, or administration of thrombolytic therapy in the last 30 days prior to randomization, or, any ECG abnormalities in the opinion of the investigator, suggestive of active ischemic changes.
* Percutaneous coronary intervention, coronary artery bypass graft surgery, other cardiac surgery, or major noncardiac surgery within 90 days prior to randomization.
* Any cardiogenic shock (SBP <90 mmHg with signs or symptoms of organ hypoperfusion) from initial presentation to randomization.
* Any significant volume depletion or severe electrolyte imbalance.
* Renal disorder with a creatinine clearance <30 mL/min, as calculated by the Cockcroft-Gault equation at screening.
* Use of a phosphodiesterase type 5 (PDE 5) inhibitor such as sildenafil within 72 hours prior to randomization.
* Planned coronary revascularization procedure (percutaneous coronary intervention or coronary artery bypass grafting) during current hospital admission.
* Use or anticipated need for invasive or noninvasive mechanical circulatory or ventilatory support.
* Anemia (hemoglobin <10 mg/dL or a hematocrit <30%).
* Vasculitis, active infective endocarditis, or suspected infections including pneumonia or sepsis.
* Body temperature ≥ 38º C.
* Significant acute or chronic respiratory disorder (eg, severe chronic obstructive pulmonary disease) or primary pulmonary hypertension with baseline dyspnea that may interfere with the ability to interpret dyspnea assessments or hemodynamic measurements.
* Terminal illness other than CHF with expected survival <180 days.
* Previous exposure to ularitide.
* Nesiritide treatment in the last 30 days prior to randomization.
* Allergy to natriuretic peptides.
* Participation in a clinical drug trial or investigational device trial within 30 days prior to randomization.
* Current drug abuse or chronic alcoholism (at the Investigator's determination).
* Women who are pregnant or breast-feeding. Women of childbearing age will have a urine pregnancy test to determine pregnancy status within 24 hours prior to randomization.
* Any condition that, in the investigator's opinion, makes the subject unsuitable for study participation, including a history of repeated admission related to non-adherence to prescribed medication.
* For subjects with concomitant invasive hemodynamic monitoring (ie, pulmonary artery catheter monitoring): Baseline PCWP ≤ 20 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)

PRIMARY OUTCOMES:
The MTD of ularitide infused over 48 hours.

SECONDARY OUTCOMES:
Frequency, severity, and relationship of AEs and serious adverse events (SAEs) to study drug through Day 32 (ie, 30 days following the end of study drug infusion).
Physical examinations, vital signs, electrocardiography, and clinical laboratory values through 48 hours.
Decline in renal function defined as a >25% rise or a 0.3 mg/dL increase in serum creatinine from pre-dose at baseline to 48 hours post the end of infusion and through Day 32.
Pharmacokinetic profile including Css, AUC, CL, V, and t½ up to 2 hours post end of infusion.
Incidence of ularitide-specific anti-drug antibodies (ADAb) through Day 32.

CONTACTS AND LOCATIONS:
Overall Officials: William Cotts, MD, Principal Investigator — Feinberg School of Medicine, Northwestern Univ.; Gregory Ewald, MD, Principal Investigator — Washington University School of Medicine; Daniel Fuleihan, MD, Principal Investigator — Cardiovascular Specialists PC dba New York Heart Ctr; Barry Greenberg, MD, Principal Investigator — UCSD Medical Center; Darshak Karia, MD, Principal Investigator — Albert Einstein Medical Center; Elie Korban, MD, Principal Investigator — Kore Cardiovascular Research Institute; Richard Nowak, MD, Principal Investigator — Henry Ford Health System; Nirav Y. Raval, MD, Principal Investigator — The Atlanta Cardiology Group, PC
Locations (8):
- United States (8):
  - UCSD Medical Center, San Diego, California
  - The Atlanta Cardiology Group, PC, Atlanta, Georgia
  - Feinberg School of Medicine, Northwestern Univ., Chicago, Illinois
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Cardiovascular Specialists PC dba New York Heart Ctr., Syracuse, New York
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Kore Cardiovascular Research Institute, Lexington, Tennessee